CLINICAL TRIAL: NCT00119080
Title: Evaluation of the Effect of Tetravalent (A, C, Y, W-135) Meningococcal Conjugate Vaccine on Serogroup-Specific Carriage of Neisseria Meningitidis
Brief Title: Effect of Meningococcal Conjugate Vaccine on Meningococcal Carriage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Georgia Department of Human Resources (Other Government); Maryland Department of Health and Mental Hygiene (Other Government); Johns Hopkins University (Other); University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCID-4591
Record Dates: First submitted 2005-07-07; First posted 2005-07-13 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Meningitis
Keywords: Meningococcal carriage; Conjugate vaccine
MeSH Terms: conditions — Meningitis | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: meningococcal conjugate vaccine (Menactra)

SUMMARY:
The purpose of this study is to determine whether the new meningococcal conjugate vaccine (MCV4) can reduce asymptomatic carriage of meningococcal bacteria, and thus decrease the transmission of these bacteria in the population.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the new meningococcal conjugate vaccine (MCV4) can reduce asymptomatic carriage of meningococcal bacteria, and thus decrease the transmission of these bacteria in the population.

Neisseria meningitidis is a leading cause of bacterial meningitis in the United States. A new tetravalent (A, C, Y, W-135) meningococcal conjugate vaccine ([MCV4], MenactraTM manufactured by Sanofi Pasteur Inc.) has been approved by Food and Drug Administration (FDA) in January 2005. This vaccine is recommended by ACIP for routine vaccination of young adolescents at the pre-adolescent visit (11-12 years old), adolescents at high school entry (15 years old), and college freshmen living in dormitories. Prevention of asymptomatic nasopharyngeal carriage of meningococci is important to interrupt person-to-person transmission and to induce herd immunity, when lower transmission results in lower disease rates among those people who are not vaccinated. No studies have yet been done to evaluate the impact of this new vaccine on carriage.

This is a randomized study designed to evaluate the effect of MCV4 on meningococcal carriage. Several high schools will be randomized into the intervention and control groups. Students in intervention group will receive MCV4 at the beginning of the study, students in the control group will be offered MCV4 after the study completion. Three specimens of throat secretions (similar to swabs for Strep throat) will be collected from the students enrolled in the study: before vaccination of intervention group students (at the start of the school year), 8 weeks post-vaccination, and 9 months post-vaccination (at the end of the school year). Questionnaire administered at the time of swabbing will assess potential risk factors for meningococcal carriage. Meningococcal bacteria isolated from the throat specimens will be serogrouped and molecularly typed. Approximately 2,000 students in each group will be needed for the study. Anticipating 35% refusal rate and 25% loss to follow-up, approximately 4,200 high school students will need to be approached in each group.

This study will answer an important question whether those who are vaccinated are protected not only from disease, but also from being asymptomatic carriers of meningococci. If so, those who are vaccinated will not be able to carry and transmit bacteria to unvaccinated individuals. Meningococcal conjugate vaccines may become available in the near future to other age groups, including infants and children. Determining the efficacy of MCV4 against meningococcal carriage will be important for policy decisions regarding vaccination with this and future conjugate vaccines in different age groups.

ELIGIBILITY:
Inclusion Criteria:

* High school students (grades 9-12) enrolled in participating schools

Exclusion Criteria:

* Contraindications to vaccine administration

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000
Dates: Start 2006-08; Study Completion 2007-05

PRIMARY OUTCOMES:
The prevalence of asymptomatic nasopharyngeal carriage of meningococci serogroup Y in vaccinated and unvaccinated individuals

SECONDARY OUTCOMES:
The overall prevalence of asymptomatic nasopharyngeal carriage of meningococci in vaccinated and unvaccinated individuals
the baseline prevalence of asymptomatic nasopharyngeal carriage of meningococci

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stern, MD, Principal Investigator — Centers for Disease Control and Prevention